CLINICAL TRIAL: NCT04284605
Title: Effects of Aerobic Training Combined With Strength Training and Yoga on Biochemical Factors, Physical Performance and Quality of Life in Patients With Pituitary Adenoma
Brief Title: Effects Exercise Training in Patients With Pituitary Adenoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra Dülger, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KA-180156
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Resistance Training; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental)
  Interventions: Other: Aerobic exercise combined with strength training; Other: Yoga
- Group2 (Experimental)
  Interventions: Other: Aerobic exercise combined with strength training; Other: Yoga

INTERVENTIONS:
Other: Aerobic exercise combined with strength training — 30 minute aerobic exercise training with warm-up and cool down followed by 30 minute strength training for specific muscles.
Other: Yoga — 60 minute yoga intervention including different asanas, breath control and meditation

SUMMARY:
This study planned to investigate the effects of aerobic training combined with strengthening training and yoga on biochemical factors, physical performance and quality of life in people with pituitary adenoma. The hypotheses are; H1: Aerobic training combined with strengthening training is effective on biochemical factors in people with pituitary adenoma.

H2: Aerobic training combined with strengthening training is effective on physical performance in people with pituitary adenoma.

H3: Aerobic training combined with strengthening training is effective on quality of life in people with pituitary adenoma.

H4: Yoga is effective on biochemical factors in people with pituitary adenoma. H5: Yoga is effective on physical performance in people with pituitary adenoma. H6: Yoga is effective on quality of life in people with pituitary adenoma. H7: Aerobic training combined with strengthening training and yoga is effective on biochemical factors, physical performance and quality of life in people with pituitary adenoma.

ELIGIBILITY:
Inclusion Criteria:

* volunteers
* macroadenomas
* at least 1 hormonal axis affected
* Karnofsky Perfomance Scale between 70-100
* 18-65 years
* approved by cardiologists

Exclusion Criteria:

* regular exercise habit
* acute pain in many part of the body
* additional neurologic condititons
* any rheumatological and immunologic conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Biochemical Factors | 6 weeks
  Concentrations of IL6, IL1beta, TNFalfa in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no IPD will be shared